CLINICAL TRIAL: NCT06185946
Title: Evaluation of Different Imaging Modalities in Regional Nodes Staging in Breast Cancer Patient
Brief Title: Evaluation of Different Imaging Modalities in Regional Lymph Nodes Staging in Patients With Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mennatallah Arous Mohamed (Other)
Responsible Party: Sponsor-Investigator, Mennatallah Arous Mohamed, assistant lecteurer, Sohag University
Organization: Sohag University (Other)
Other Study IDs: Soh_med_23_11_02MD
Record Dates: First submitted 2023-11-29; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Breast Carcinoma Metastatic in Lymph Node

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ultrasonography group
- mammoragraphy group: patient with ultrasoundy only
- CT group: pateint with postive node undergo further staging
- MRI group: patient whit postive node with staging

SUMMARY:
The regional lymph node status is considered to be an important prognostic factor regarding the long-term survival of breast cancer (BC) patients (Cetin IA, et al . 2020). The knowledge of whether lymph nodes are tumor-infiltrated or not is essential since nodal involvement has decisive therapeutic consequences such as axillary lymph node dissection (ALND), axillary radiotherapy, and neoadjuvant or adjuvant systemic chemotherapy (Diessner J et al . 2023). To provide individualized therapeutic options and optimized therapy.

DETAILED DESCRIPTION:
The following data will be collected from electronic or paper medical data records as:

1) Age 2 )Sex 3)Family history of breast cancer 4)Menopausal status 5 )Body mass index (BMI) 6) Histological type of BC as reported in pathology 7) The results of the lymph node status. 8)Registered data will be collected from the hospital databases and clinical sheers. 3 9) The gold standard reference in the evaluation of suspicious lymph nodes by nodal biopsy and postoperative pathology. Imaging technique and interpretation The imaging diagnostic for BC (MRI, CT, mammography, and ultrasound) patients are carried out by the Department of Diagnostic and Interventional Radiology of the Hospitals in the research and interpreted by radiologists at the time of BC diagnosis. The radiological reports for each patient and each imaging technique will be analyzed about the lymph node status. The nodal status will be reported as benign, indeterminate, and infiltrated as stated by the ACR lexicon. Mammography and US For mammography, we will use full-field digital mammography systems with the option of additional tomosynthesis for further characterization of the primary tumor at NCI with the commercially available The BC patients routinely receive an ultrasound exam including the evaluation of the breast and the axilla with the lymphatic drainage pathways as a part of the follow-up process active lymph nodes. p values lower than 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patient consenting to participate in the study.
2. Patients who can tolerate the imaging modalities and have proven to tolerate the contrast agents . 3) Breast cancer patients coming for an initial assessment with or without clinical regional lymph nodes positive status.

4) Breast cancer patients planned to have(breast-conserving surgery or mastectomy)as well as lymph node surgeries(sentinel lymph node v biopsy and/or axillary lymph node dissection.

Exclusion Criteria:

1)Patients denying consent to participate in the study 2) Patients who are not fit for further imaging evaluation (patients who exceed the weight limit, patients who are sensitive to contrast material, etc). 3) Patients with bilateral MRM and AC

-

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female over 25 years
Study Population: The plan is to study a population of 100 patients of BC presenting to Sohag university And NCI in breast cancer clinic surgery the Late 2023 and 2024
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-12 (Estimated)

PRIMARY OUTCOMES:
evaluate the sensitivity of different Imaging modality pretherapeutic imaging modalities (sonography, mammography, CT and MRI) in pretherapeutic assessment of nodal-status in BC patients . | one year

SECONDARY OUTCOMES:
to find out if there is further benefit of using cross-sectional imaging (MRI, CT) for pretherapeutic axillary staging compared to Us and mammogram conventional imaging such as mammography and sonogram. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Hattali S, Vinnicombe SJ, Gowdh NM, Evans A, Armstrong S, Adamson D, Purdie CA, Macaskill EJ. Breast MRI and tumour biology predict axillary lymph node response to neoadjuvant chemotherapy for breast cancer. Cancer Imaging. 2019 Dec 26;19(1):91. doi: 10.1186/s40644-019-0279-4. PMID 31878958
- [Background] Bakker MF, de Lange SV, Pijnappel RM, Mann RM, Peeters PHM, Monninkhof EM, Emaus MJ, Loo CE, Bisschops RHC, Lobbes MBI, de Jong MDF, Duvivier KM, Veltman J, Karssemeijer N, de Koning HJ, van Diest PJ, Mali WPTM, van den Bosch MAAJ, Veldhuis WB, van Gils CH; DENSE Trial Study Group. Supplemental MRI Screening for Women with Extremely Dense Breast Tissue. N Engl J Med. 2019 Nov 28;381(22):2091-2102. doi: 10.1056/NEJMoa1903986. PMID 31774954
- [Background] Caudle AS, Yang WT, Krishnamurthy S, Mittendorf EA, Black DM, Gilcrease MZ, Bedrosian I, Hobbs BP, DeSnyder SM, Hwang RF, Adrada BE, Shaitelman SF, Chavez-MacGregor M, Smith BD, Candelaria RP, Babiera GV, Dogan BE, Santiago L, Hunt KK, Kuerer HM. Improved Axillary Evaluation Following Neoadjuvant Therapy for Patients With Node-Positive Breast Cancer Using Selective Evaluation of Clipped Nodes: Implementation of Targeted Axillary Dissection. J Clin Oncol. 2016 Apr 1;34(10):1072-8. doi: 10.1200/JCO.2015.64.0094. Epub 2016 Jan 25. PMID 26811528
- [Background] Cetin IA, Akay SU, Caglar Ozkok HB, Sengoz M. Lymph node ratio as an independent prognostic factor for breast cancer-related mortality in patients with node-positive breast cancer. J Cancer Res Ther. 2020 Oct-Dec;16(6):1387-1392. doi: 10.4103/jcrt.JCRT_1034_19. PMID 33342802
- [Background] Choi HY, Park M, Seo M, Song E, Shin SY, Sohn YM. Preoperative Axillary Lymph Node Evaluation in Breast Cancer: Current Issues and Literature Review. Ultrasound Q. 2017 Mar;33(1):6-14. doi: 10.1097/RUQ.0000000000000277. PMID 28187012
- [Background] de Meric de Bellefon M, Lemanski C, Ducteil A, Fenoglietto P, Azria D, Bourgier C. Management of the Axilla in the Era of Breast Cancer Heterogeneity. Front Oncol. 2018 Apr 4;8:84. doi: 10.3389/fonc.2018.00084. eCollection 2018. PMID 29670853
- [Background] Diessner J, Anders L, Herbert S, Kiesel M, Bley T, Schlaiss T, Sauer S, Wockel A, Bartmann C. Evaluation of different imaging modalities for axillary lymph node staging in breast cancer patients to provide a personalized and optimized therapy algorithm. J Cancer Res Clin Oncol. 2023 Jul;149(7):3457-3467. doi: 10.1007/s00432-022-04221-9. Epub 2022 Aug 10. PMID 35948829
- [Background] Ditsch N, Untch M, Kolberg-Liedtke C, Jackisch C, Krug D, Friedrich M, Janni W, Muller V, Albert US, Banys-Paluchowski M, Bauerfeind I, Blohmer JU, Budach W, Dall P, Diel I, Fallenberg EM, Fasching PA, Fehm T, Gerber B, Gluz O, Hanf V, Harbeck N, Heil J, Huober J, Kreipe HH, Kuhn T, Kummel S, Loibl S, Luftner D, Lux M, Maass N, Moebus V, Mundhenke C, Park-Simon TW, Reimer T, Rhiem K, Rody A, Schmidt M, Schneeweiss A, Solbach C, Solomayer EF, Stickeler E, Thomssen C, Witzel I, Wockel A, Thill M. AGO Recommendations for the Diagnosis and Treatment of Patients with Locally Advanced and Metastatic Breast Cancer: Update 2020. Breast Care (Basel). 2020 Jun;15(3):294-309. doi: 10.1159/000508736. Epub 2020 Jun 10. No abstract available. PMID 32774225
- [Background] Dong Y, Feng Q, Yang W, Lu Z, Deng C, Zhang L, Lian Z, Liu J, Luo X, Pei S, Mo X, Huang W, Liang C, Zhang B, Zhang S. Preoperative prediction of sentinel lymph node metastasis in breast cancer based on radiomics of T2-weighted fat-suppression and diffusion-weighted MRI. Eur Radiol. 2018 Feb;28(2):582-591. doi: 10.1007/s00330-017-5005-7. Epub 2017 Aug 21. PMID 28828635
- [Background] El Sabbagh YH, Hamdy O. Targeted Axillary Dissection In Breast Cancer Patients After Neoadjuvant Therapy. Mansoura Medical Journal. 2022 Dec 1;51(4):246-57.
- [Background] Johnston SRD, Harbeck N, Hegg R, Toi M, Martin M, Shao ZM, Zhang QY, Martinez Rodriguez JL, Campone M, Hamilton E, Sohn J, Guarneri V, Okada M, Boyle F, Neven P, Cortes J, Huober J, Wardley A, Tolaney SM, Cicin I, Smith IC, Frenzel M, Headley D, Wei R, San Antonio B, Hulstijn M, Cox J, O'Shaughnessy J, Rastogi P; monarchE Committee Members and Investigators. Abemaciclib Combined With Endocrine Therapy for the Adjuvant Treatment of HR+, HER2-, Node-Positive, High-Risk, Early Breast Cancer (monarchE). J Clin Oncol. 2020 Dec 1;38(34):3987-3998. doi: 10.1200/JCO.20.02514. Epub 2020 Sep 20. PMID 32954927
- [Background] Kutomi G, Ohmura T, Satomi F, Takamaru T, Shima H, Suzuki Y, Otokozawa S, Zembutsu H, Mori M, Hirata K. Lymph node shape in computed tomography imaging as a predictor for axillary lymph node metastasis in patients with breast cancer. Exp Ther Med. 2014 Aug;8(2):681-685. doi: 10.3892/etm.2014.1787. Epub 2014 Jun 16. PMID 25009640
- [Background] Lee SC, Jain PA, Jethwa SC, Tripathy D, Yamashita MW. Radiologist's role in breast cancer staging: providing key information for clinicians. Radiographics. 2014 Mar-Apr;34(2):330-42. doi: 10.1148/rg.342135071. PMID 24617682
- [Background] Marino MA, Avendano D, Zapata P, Riedl CC, Pinker K. Lymph Node Imaging in Patients with Primary Breast Cancer: Concurrent Diagnostic Tools. Oncologist. 2020 Feb;25(2):e231-e242. doi: 10.1634/theoncologist.2019-0427. Epub 2019 Oct 14. PMID 32043792
- [Background] Masuda N, Lee SJ, Ohtani S, Im YH, Lee ES, Yokota I, Kuroi K, Im SA, Park BW, Kim SB, Yanagita Y, Ohno S, Takao S, Aogi K, Iwata H, Jeong J, Kim A, Park KH, Sasano H, Ohashi Y, Toi M. Adjuvant Capecitabine for Breast Cancer after Preoperative Chemotherapy. N Engl J Med. 2017 Jun 1;376(22):2147-2159. doi: 10.1056/NEJMoa1612645. PMID 28564564
- [Background] Shirzadi A, Mahmoodzadeh H, Qorbani M. Assessment of sentinel lymph node biopsy after neoadjuvant chemotherapy for breast cancer in two subgroups: Initially node negative and node positive converted to node negative - A systemic review and meta-analysis. J Res Med Sci. 2019 Feb 25;24:18. doi: 10.4103/jrms.JRMS_127_18. eCollection 2019. PMID 30988686
- [Background] Telli ML, Gradishar WJ, Ward JH. NCCN Guidelines Updates: Breast Cancer. J Natl Compr Canc Netw. 2019 May 1;17(5.5):552-555. doi: 10.6004/jnccn.2019.5006. PMID 31117035
- [Background] von Minckwitz G, Huang CS, Mano MS, Loibl S, Mamounas EP, Untch M, Wolmark N, Rastogi P, Schneeweiss A, Redondo A, Fischer HH, Jacot W, Conlin AK, Arce-Salinas C, Wapnir IL, Jackisch C, DiGiovanna MP, Fasching PA, Crown JP, Wulfing P, Shao Z, Rota Caremoli E, Wu H, Lam LH, Tesarowski D, Smitt M, Douthwaite H, Singel SM, Geyer CE Jr; KATHERINE Investigators. Trastuzumab Emtansine for Residual Invasive HER2-Positive Breast Cancer. N Engl J Med. 2019 Feb 14;380(7):617-628. doi: 10.1056/NEJMoa1814017. Epub 2018 Dec 5. PMID 30516102